CLINICAL TRIAL: NCT00495833
Title: SPHERE Hypertension Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Hendrika Meischke, Professor, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: 32168-E/G; 07-6656-E/G 01
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 1 (No Intervention)
- 2 (Experimental): photo and blood pressure personalization
  Interventions: Behavioral: Personalized brochure
- 3 (Experimental): photo personalization only
  Interventions: Behavioral: Personalized brochure
- 4 (Experimental): blood pressure personalization only
  Interventions: Behavioral: Personalized brochure
- 5 (Experimental): no personalization
  Interventions: Behavioral: Personalized brochure
- A (Experimental): receives gift card in blood pressure (BP) kit
  Interventions: Behavioral: Promotional gift
- B (Experimental): does not receive gift card in BP kit
  Interventions: Behavioral: Promotional gift

INTERVENTIONS:
Behavioral: Personalized brochure — either photo personalization, blood pressure personalization, both, or no personalization
  Arms: 2; 3; 4; 5
Behavioral: Promotional gift — half of participants who go to a fire station will receive a gift card.
  Arms: A; B

SUMMARY:
Overview: This study uses communications strategies delivered through the traditional emergency medical response system to increase the proportion of low-income adults who obtain blood pressure screening and follow-up information for hypertension treatment options. The project will test the effectiveness of source personalization and tailored messaging in motivating potentially high-risk people, identified by 911 responders, to come to a local fire station for hypertension screening.

Specific Aims: The specific aims are:

1. Test the effectiveness of three health marketing approaches to motivate high-risk people, identified via 911 responders, to come to a local fire station for hypertension screening. The mailed marketing approaches vary personalized risk information and personalization of source.
2. Test the effectiveness of two mailing interventions (blood pressure kits with and without promotional gifts) to increase blood pressure monitoring among patients who have come to a fire station for a second blood pressure check.

DETAILED DESCRIPTION:
Hypertension, if left untreated, is a major risk factor for stroke, heart attack, heart failure or kidney failure. Many people with hypertension don't know they have the disease and/or may be under treated. As such they are at higher risk for health complications than those who are managing their condition.

People who see a regular healthcare provider are more likely to know they have hypertension, and they are more likely to receive appropriate treatment. However, many patients who call 9-1-1 for emergency medical services (EMS) do not have regular health care providers and may be more at risk for undiagnosed or under treated disease.

EMS personnel enter the homes of thousands of residents each year. Emergency medical technicians (EMTs) routinely take patients' blood pressure as part of their standard diagnostic procedures. EMTs and paramedics complete a medical incident report form (MIRF) for each patient, including this information. As recorded on the MIRFs, thousands of patients have high blood pressure (defined by a systolic measurement of 160 or higher and/or a diastolic measurement of 100 or higher) during those visits. Blood pressure may be elevated simply from the stress and anxiety of a 9-1-1 response. But even in light of this potential "white coat" phenomenon, blood pressure readings at these levels are very high and are a cause for concern, especially in cases where patients are not transported to the hospital for further examination.

From February - April, 2007 we are collecting baseline data on patients who have high blood pressure readings (160/100 or higher) at a 9-1-1 response by an EMT (SPHERE Hypertension Baseline Data Study). We want to understand what these patients remember during the 9-1-1 response around their high blood pressure measure, if the patients seek a second reading, and if the patients seek follow-up care as a result of the high blood pressure measure. We are also interested to learn if patients trust EMTs as a provider of preventive health care. This baseline data will also allow us to more accurately measure the success of this proposed intervention study. The baseline data collection is almost completed and we now will proceed with an intervention study.

We propose to conduct an intervention study next, aimed at:

* Motivating subjects to receive a follow-up hypertension assessment from an EMT at a local fire station after receiving a high blood pressure reading from an EMT during a 911 event.
* Motivating subjects to monitor their blood pressure as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Seen by EMTs in one of the four participating fire departments (Bellevue, Kent, Renton, Shoreline)
* Recorded systolic blood pressure >= 160 and/or diastolic blood pressure >= 100
* At least 18 years old

Exclusion Criteria:

* Patient transported by paramedics
* Patient nursing home/adult family home resident
* Patient a prisoner or in custody (in jail or at the Regional Justice Center in Kent, for example)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The effectiveness of three health marketing approaches to motivate high-risk people, identified via 911 responders, to come to a local fire station for hypertension screening. | June 2007-June 2009
The effectiveness of two mailing interventions (blood pressure kits with and without promotional gifts) to increase blood pressure monitoring among patients who have come to a fire station for a second blood pressure check. | June 2007 - June 2009

SECONDARY OUTCOMES:
Test if non-responders have lower trust in, and/or lower perceived efficacy of, the fire stations as preventive health care providers than participants who go to the fire station for a blood pressure check. | June 2007 - December 2009
Correlate the resulting health behaviors with existing health disparity indicators (including health literacy, socioeconomic status, and rural residence) | June 2007 - December 2009
Cost analysis | June 2007 - December 2009

CONTACTS AND LOCATIONS:
Overall Officials: Hendrika Meischke, PhD, Principal Investigator — University of Washington; Mickey Eisenberg, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Health Promotion Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Meischke H, Ike BR, Fahrenbruch C, Kuniyuki A, Hannon P, Parks MR, Forehand M, Weaver M, Harris JR. Hypertension identification via emergency responders: a randomized controlled intervention study. Prev Med. 2013 Dec;57(6):914-9. doi: 10.1016/j.ypmed.2013.05.010. Epub 2013 Jun 1. PMID 23732250